CLINICAL TRIAL: NCT05299775
Title: Poor Quality of Life Associated With Traditional Chinese Medicine Constitution in HIV-infected Men Who Have Sex With Men
Status: Completed | Type: Observational
Sponsor: Taipei City Hospital (Other Government)
Responsible Party: Principal Investigator, Chung-Hua Hsu, Clinical professor, Taipei City Hospital
Other Study IDs: TCHIRB-10707110
Record Dates: First submitted 2021-12-08; First posted 2022-03-29 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: HIV Infections; Quality of Life
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HIV infected time: Group are divided by Infected time: 0-2W, 2W-12M, >1Y
  Interventions: Diagnostic Test: World Health Organization Quality of Life -Brief -Taiwan version (WHOQOL-BREF-Taiwan version)
- different constitutions: Group are divided by different constitutions:It includes 9 basic types of constitution, yang deficiency , yin deficiency , qi deficiency , phlegm dampness , damp-heat, blood stasis, special diathesis , qi depression , gentleness constitution .

INTERVENTIONS:
Diagnostic Test: World Health Organization Quality of Life -Brief -Taiwan version (WHOQOL-BREF-Taiwan version) — WHOQOL-BREF-Taiwan version is used to measure the quality of life in HIV infected.
  Wang Qi nine kinds of TCM constitution Questionnaire is used to measure the constitution of HIV infected.
  Other Names: Wang Qi nine kinds of TCM constitution Questionnaire
  Groups: HIV infected time

SUMMARY:
This study explores the pathological constitution as it relates to low quality of life with HIV- infected MSM patients, as a reference for clinical treatment.

DETAILED DESCRIPTION:
Introduction :This study explores the pathological constitution as it relates to low quality of life with HIV- infected MSM patients, as a reference for clinical treatment.

Methods :It has a cross-sectional research design using structured questionnaires to collect data,including patient's basic case data, CD4+, CD4+/CD8+ ratio, Wang Qi constitution and WHOQOL-BREF -Taiwan version questionnaires. We consider the association between the constitutions and quality of life for HIV-infected MSM patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with HIV infected.
* Age greater than 20 years old (including) and less than 60 years old.
* Conscious clear and voluntary to attend the project with agreement.
* Willing to fill out the informed consent form.

Exclusion Criteria:

* conscious unclear
* Patients had histories of severe psychiatric disorders ( ex: schizophrenia) or if they met the criteria of Diagnostic and Statistical Manual of Mental Disorders ( ex: dementia)
* Age < 20 years old.
* The patient does not want to fill out the informed consent form for any reason.

Ages: 20 Years to 49 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Study Population: We invited all people diagnosed with HIV infected through MSM in the outpatient Department of Infection, Taipei City United Hospital, Linsen Chinese Medicine and Kunming Branch, to participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 203 (Actual)
Dates: Start 2018-09-21 (Actual); Primary Completion 2019-02-18 (Actual); Study Completion 2019-07-09 (Actual)

PRIMARY OUTCOMES:
quality of life score | Lasts for 1 year
  investigate different quality of life score of HIV infected time in the physical,psychological, social, and environmental domains.
  Outcome Measure:4 quality of life scores for each constitution ， In the WHOQOL-BREF Taiwan item scores range from 1 (worst condition) to 5 (best condition), except for 3 items (Ph1, Ph2, and Ps6), which have reverse scores. Two scales (0-100 and 4-20, with a higher score indicating better QOL) can be transformed into domain scores for each domain and we used the 4-20 scale in this study,Add the item scores for each domain ,the higher scores indicating better quality of life
TCM constitution | Lasts for 1 year
  Investigate TCM constitution composed of HIV-infected in yang deficiency , yin deficiency , qi deficiency , phlegm dampness , damp-heat , blood stasis , special diathesis , qi stagnation , and gentleness constitution .
  Outcome Measure:Nine kinds TCM constitution-the constitution type must be judged according to the standards. Original score = sum of the scores of items for each constitution, and then the original score is converted into a conversion score [conversion score = [(original score-number of answer items) / answer items × 4] × 100.
  Judgment of constitutions: gentleness is a normal constitution, and others are pathological constitutions. Gentleness constitution conversion score ≥ 60 points, and other pathological constitution conversion score <30 points, it is Gentleness constitution; pathological constitution conversion score ≥ 40 is considered pathological constitution, The higher the conversion score is the more obvious the constitution trend

CONTACTS AND LOCATIONS:
Overall Officials: Chung-Hua Hsu, Study Director — clinical professor
Locations (1):
- Taipei City Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided